CLINICAL TRIAL: NCT04706455
Title: Effect of Artificial Tears on the Parameters of the Eye in Normal and Dry Eyes and Its Impact on IOL Power Calculation for Cataract Surgery
Brief Title: Effect of Artificial Tears on the Parameters of the Eye and Its Impact on IOL Power Calculation for Cataract Surgery
Acronym: IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20210312
Record Dates: First submitted 2020-12-20; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Cataract Senile; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Corneal topography and Biometry will be performed in individuals with age-relate cataract. Patients will be classified as dry eye or normal eye based on BUT. The tear film breakup (BUT) time of less than 5 seconds will be diagnosed as dry eyes. One of two artificial tear eye drops will be instilled in the eye, and corneal topography and biometry will be repeated after 5 minutes of application
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium hyaluronate 0.1% (Active Comparator): First preoperative Biometry of the eye at the IOL Master® will be measured. Then, corneal topography will be measure at the Oculus pentacam®. Afterwards, sodium hyaluronate 0.1% will be installed and biometry and corneal topography will be repeated after 5 minutes.
  Interventions: Device: sodium hyaluronate 0.1%
- sodium hyaluronate 0.3% (Active Comparator): First preoperative Biometry of the eye at the IOL Master® will be measured. Then,corneal topography will be measure at the Oculus pentacam®. Afterwards, sodium hyaluronate 0.3% will be installed and biometry and corneal topography will be repeated after 5 minutes.
  Interventions: Device: sodium hyaluronate 0.3%

INTERVENTIONS:
Device: sodium hyaluronate 0.1% — Instillation of one drop sodium hyaluronate 0.1%
  Arms: sodium hyaluronate 0.1%
Device: sodium hyaluronate 0.3% — Instillation of one drop sodium hyaluronate 0.3%
  Arms: sodium hyaluronate 0.3%

SUMMARY:
First, preoperative biometry of the eye at the IOL Master® will be performed. Then, corneal topography will be measured at the Oculus pentacam®. Afterwards, one of two eye drops are instilled in the eye, and biometry and corneal topography will be repeated after 5 minutes.

For all patients, the Barrett Universal II formula will be used for calculation of IOL power. Predicted refraction outcome will be referred to as SEQ. The chief surgeon will perform the uneventful standard cataract operation with in-the-bag implantation of a HOYA IOL (Model 251) through a 2.4-mm corneal incision.

A Subjective Refraction using plus principle will be performed one month after the operation, and ETDRS visual acuity charts will be used to measure best-corrected visual acuity. Refraction will be described as SR (postoperative SEQ) and will be calculated as:

SR = sphere + (0.5*cylinder)

DETAILED DESCRIPTION:
First, preoperative biometry of the eye at the IOL Master® will be performed. Then, corneal topography will be measured at the Oculus pentacam®. Patients will be classified as dry eye or normal eye based on BUT. The tear film breakup (BUT) time of less than 5 seconds will be diagnosed as dry eyes.Afterwards, one of two eye drops are instilled in the eye, and biometry and corneal topography will be repeated after 5 minutes.

For all patients, the Barrett Universal II formula will be used for calculation of IOL power. Predicted refraction outcome will be referred to as SEQ. The chief surgeon will perform the uneventful standard cataract operation with in-the-bag implantation of a HOYA IOL (Model 251) through a 2.4-mm corneal incision.

A Subjective Refraction using plus principle will be performed one month after the operation, and ETDRS visual acuity charts will be used to measure best-corrected visual acuity. Refraction will be described as SR (postoperative SEQ) and will be calculated as:

SR = sphere + (0.5*cylinder)

ELIGIBILITY:
Inclusion Criteria:

* A patient diagnosed with age related cataract
* 30 to 95 years old
* Medical history and physical examination should be normal.

Exclusion Criteria:

* • Abnormality of the cornea (scaring of the cornea)

  * If any topical therapy (i.e. glaucoma) of the eye is needed
  * Active allergy of eye or nose
  * Any conjunctivitis or keratitis
  * If nasolacrimal drainage apparatus is abnormal
  * severity level 4 of dry eye (constant discomfort in the eye accompanied with visual symptoms, filamentary keratitis, , keratinization, severe conjunctival injection, ulceration clumping of mucus glands, tear debris, , trichiasis, symblepharon)
  * deformities of lid
  * Preceding eye trauma or surgery
  * Any Uncontrolled ocular disease or systemic disease
  * Lactation
  * Pregnancy

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
keratometric value of the eye measured with Master 500 before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  k-value (k, k1, k2 in Diopter)
Axial length of the eye measured with Master 500 before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  Axial length (AL in mm)
Anterior chamber depth of the eye measured with Master 500 before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  Anterior chamber depth (ACD in mm)
Sim K of the eye measured with Oculus Pentacam before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  Sim K (k1, k2 in Diopter)
Total Corneal Refractive Power of the eye measured with Oculus Pentacam before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  Total Corneal Refractive Power (TCRP in Diopter),
Total Corneal Irregular Astigmatism of the eye measured with Oculus Pentacam before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  Total Corneal Irregular Astigmatism (TCIA in Diopter)
Predicted spherical equivalent (SE) calculated with Barrett Universal II formula before and after 5 minutes of installation of artificial tears (sodium hyaluronate 0.1% or 0.3% eye drops). | 5 minutes
  Predicted spherical equivalent (SEQ in Diopter)
Postoperative spherical equivalent (SE) measured one month after surgery. | one month after surgery
  Postoperative spherical equivalent (SE in Diopters)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Bai, MD,PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Department of Ophthalmology, Second affiliated hospital of Xian Jiaotong University, Xi'an, Shaanxi, China